CLINICAL TRIAL: NCT00359359
Title: Phase I/II Study to Investigate the Safety, Tolerability, Efficacy and Pharmacokinetics of ZK 219477 in Combination With Cisplatin as First-line Therapy in Chemotherapy-naïve Patients With Extensive-disease (ED) Stage Small-cell Lung Cancer (SCLC)
Brief Title: A Study of a New Chemotherapy Agent in Combination With Cisplatin to Treat Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91495; 2006-000067-29 (EudraCT Number); 310101 (Other: Company Internal)
Record Dates: First submitted 2006-07-27; First posted 2006-08-02 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoma, Small Cell
Keywords: Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma | interventions — sagopilone; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sagopilone and cisplatin (Experimental): The study drug sagopilone was administered in combination with a fixed dose of cisplatin
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477); Drug: Cisplatin

INTERVENTIONS:
Drug: Sagopilone (BAY86-5302, ZK 219477) — Phase 1: dose escalation/deescalation, starting dose 12mg/m² Sagopilone, Phase 2: MTD or RPIID
Drug: Cisplatin — 75 mg/m² as a 1 h infusion after the sagopilone infusion on Day 1

SUMMARY:
The purpose of the study is to determine whether the study drug ZK 219477 (also known as SH Y03757A) combined with cisplatin, is effective in the treatment of small cell lung cancer in patients who did not receive prior treatment for their lung cancer

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Small-cell lung cancer
* Stage of extensive disease
* Adequate function of major organs and systems
* Use of highly effective birth control methods in females of child-bearing potential

Exclusion Criteria:

* Prior chemotherapy for small-cell lung cancer
* Prior surgical resection or radiotherapy for SCLC within at least 3 to 4 weeks prior to inclusion and with the exception of radiation of brain metastases
* Superior vena cava syndrome or obstruction of any vital structure
* Untreated malignant hypercalcemia; Extensive disease amenable to radiation therapy; Symptomatic brain metastases requiring whole-brain irradiation
* Known allergy or hypersensitivity to platinum-containing drugs
* Pregnancy or breast-feeding
* Use of any investigational drug within 4 weeks before start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety measure to establish the MTD or RPDII dose of Sagopilone used in combination with cisplatin | Phase 1: Baseline up to 3 month of treatment
Phase 2: Efficacy measure | Phase 2: every 6 weeks after start of treatment

SECONDARY OUTCOMES:
Phase 1: PK of Sagopilone + Cisplatin | Upto 336 h after the beginning of the sagopilone infusion and upto 20 h 45 min after the beginning of the cisplatin infusion
Phase 2: Duration of CR or PR | every 6 weeks after start of treatment
  Duration of complete response (CR) or partial response (PR) as 'overall response', defined as time between first date that the measurement criteria for CR or PR as 'overall response' are met and first date that recurrence or overall response of (progressive disease) PD is documented.
Phase 2: TTP | every 6 weeks after start of treatment
  Time to tumor progression (TTP) is defined as the time from the date of treatment assignment to the first observation of disease progression or to the last date of a definite assessment (not status unknown), if the patient is progression-free until that assessment.
Phase 2: PFS | every 6 weeks after start of treatment
  Progression free survival (PFS) is defined as the time from date of treatment assignment to the first observation of disease progression or death of any cause or to the last date of a definite assessment (not status unknown), if the patient was progression-free until that assessment
Phase 2: OS | every 3 months after start of treatment
  Overall survival (OS) is defined as the time from date of treatment assignment until death from any cause or until the last date the patient is known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Germany (9):
  - Gerlingen, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - München, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Wiesbaden, Hesse
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Berlin, State of Berlin